CLINICAL TRIAL: NCT07159269
Title: Cardiac Point-of-care Ultrasound Clinical Training Pathway Implementation and Impact Assessment for Advanced Practice Providers in the Emergency Department
Brief Title: Cardiac point-of Care Ultrasound Training Pathway for Emergency Department Advanced Practice Providers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00118464
Record Dates: First submitted 2025-08-20; First posted 2025-09-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Disease Acute; Emergency Department Patient; Heart Failure Acute; Pulmonary Embolism (Diagnosis); Point of Care Ultrasound (POCUS); Cardiac Tamponade; Pericardial Effusion; Diagnostic Imaging; Medical Training; Implementation Science
Keywords: point of care ultrasound; focused cardiac ultrasound; advanced practice provider training; medical education; implementation science
MeSH Terms: conditions — Pulmonary Embolism; Disease; Cardiac Tamponade; Pericardial Effusion | interventions — Critical Pathways

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced Practice Provider (APP) Cohort (Experimental): Advanced Practice Providers (APPs) are nonphysicians essential to the emergency department workforce, especially in rural and community hospitals.
  Interventions: Behavioral: Cardiac point-of-care ultrasound (POCUS) training and clinical pathway

INTERVENTIONS:
Behavioral: Cardiac point-of-care ultrasound (POCUS) training and clinical pathway — Participants will complete a cardiac POCUS simulation session and a hands-on observed structured clinical skill exam (OSCE) post-training led by ultrasound-trained faculty. Then as part of standard clinical care, advanced practice providers (APPs) will perform POCUS while supervised by emergency medicine (EM) attending physicians. To assess program feasibility and acceptability, participants will complete a pre/post and 6-month post-survey and semi-structured interview, as well as a knowledge and technical skills assessment.

SUMMARY:
The aim of this study is to assess emergency medicine physician and advanced practice provider (APP) knowledge and technical skill in performance of a point-of-care ultrasound simulation and just-in-time training pathway to determine the feasibility, acceptability, and usability of the ultrasound training program. By performing this study, we hope to create a standardized training model which could potentially facilitate point-of-care ultrasound (POCUS) clinical performance and thereby improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* advanced practice providers (APPs) currently working in our ED, with additional APPs as they are hired (expected to be about 75 APPs total within the next 3 years due to expanding staffing needs and coverage models).

Exclusion Criteria:

* non-APPs such as physicians, nurses, or other clinical staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Assess the feasibility of implementing a just-in-time cardiac point-of-care ultrasound (POCUS) clinical training pathway for advanced practice providers (APPs) using the Reach Effectiveness Adoption Implementation Maintenance (RE-AIM) framework. | 1-2 years for each study site
  Participants will complete a cardiac POCUS simulation session and a hands-on structured clinical skill exam post-training (OSCE) led by ultrasound-trained faculty. Then as part of standard clinical care, APPs will perform POCUS while supervised by EM attending physicians. The primary outcome assesses program feasibility and acceptability. Participants will complete a pre/post and 6-month post-survey and semi-structured interview. Survey questions are structured based on the Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) survey tool. This is scored on a Likert scale from 1-5.
Aim 1: Acceptability of the Intervention as measured by the Acceptability of Intervention Measure (AIM) | 1-2 years for each study site
  The AIM is scored on a Likert scale from 1 to 5, where a higher score indicates greater acceptability.
Aim 1: Appropriateness of the Intervention as measured by the Intervention Appropriateness Measure (IAM) | 1-2 years for each study site
  The IAM is scored on a Likert scale from 1 to 5, where a higher score indicates greater appropriateness.
Aim 1: Feasibility of the Intervention as measured by the Feasibility of Intervention Measure (FIM) survey tool | 1-2 years for each study site
  The FIM is scored on a Likert scale from 1 to 5, where a higher score indicates greater appropriateness.

SECONDARY OUTCOMES:
Aim 1: Feasibility of implementing a just-in-time cardiac point-of-care ultrasound (POCUS) clinical training pathway for advanced practice providers (APPs) using the Reach Effectiveness Adoption Implementation Maintenance (RE-AIM) framework. | 1-2 years for each study site
  Using a modified framework analysis approach, a team of 3-4 trained research assistants and the two emergency ultrasound fellows led by an implementation science expert will deductively analyze semi-structured interview content based on RE-AIM constructs with open inductive coding for data that does not fit into the framework. The investigators will perform a preliminary rapid qualitative deductive analysis based on audio recordings and meeting notes applied to the RE-AIM dimensions, to determine scope and saturation. Coding and categorization will be conducted with RE-AIM templated coding sheets and transferred to NVivo.
Aim 2: Educational impact of the training model on point-of-care ultrasound (POCUS) use and diagnostic performance | 1-2 years for each study site
  Participants will complete a pre-, post-, and 6-month post-training knowledge assessment and technical skill test to assess the educational impact of the cardiac POCUS program, structured using the Ultrasound Competency Assessment Tool (UCAT), which is scored on a Likert scale from 1-5, where a higher score indicates greater competency.
Aim 2: Clinical impact of the training model on point-of-care ultrasound (POCUS) use and diagnostic performance - number of clinical POCUSs performed | 1-2 years for each study site
  To assess the advanced practice provider (APP) training program effectiveness, the investigators will collect pre/post-health record data on the number of clinical POCUS performed in the emergency department pre/post-intervention (from the Butterfly ultrasound archiving system, units in counts/percentages).
Aim 2: Clinical impact of the training model on point-of-care ultrasound (POCUS) use and diagnostic performance - image quality | 1-2 years for each study site
  To assess APP training program effectiveness, the investigators will collect pre/post-health record data on image quality review scores (determine by two ultrasound experts, Likert scale 1-5, where a higher score indicates greater quality).
Aim 2: Clinical impact of the training model on point-of-care ultrasound (POCUS) use and diagnostic performance - diagnostic accuracy | 1-2 years for each study site
  The investigators will collect data on diagnostic accuracy as compared to radiology studies (from ultrasound expert review, True Positive, True Negative, False Positive, False Negative, or Technically-limited study)
Aim 2: Clinical impact of the training model on point-of-care ultrasound (POCUS) use and diagnostic performance - time to initial cardiology consult | 1-2 years for each study site
  The investigators will collect electronic health record data on pre/post-intervention time to initial cardiology consult (both from the Epic electronic health record, units in hours).
Aim 2: Clinical impact of the training model on point-of-care ultrasound (POCUS) use and diagnostic performance - emergency department length-of-stay | 1-2 years for each study site
  The investigators will collect electronic health record data on pre/post-intervention ED length-of-stay (from the Epic electronic health record, units in hours).
Aim 2: Impact of the training model on cost-effectiveness | 1-2 years for each study site
  The investigators will collect pre/post-intervention POCUS revenue data for cost-effectiveness (from hospital billing data, units in dollars).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca G Theophanous, MD, MHSc, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No